CLINICAL TRIAL: NCT02839395
Title: The Effects of Acute vs. Chronic of Screen Illumination on: Sleep Efficacy and Architecture, Physiology, Emotion and Behavior: Possible Effect on Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Lilach Kemer, Dr., Assuta Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 0005-16-ASMC
Record Dates: First submitted 2016-07-07; First posted 2016-07-21 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Sleep; Emotion
Keywords: screen illumination; melatonin; body temperature; cognitive functioning; light pollution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- base line (Active Comparator): First night is the base line- no exposure to computer screen illumination.
  Interventions: Other: No intervention- base line
- Acute (Experimental): Second night is the acute exposure to computer screen illumination.
  Interventions: Other: Acute
- Chronic (Experimental): Chronic is the effect after five nights of exposure to computer screen light illumination.
  Interventions: Other: Chronic

INTERVENTIONS:
Other: No intervention- base line — the subject will sited in a dim light room. No screen light illumination.
  Arms: base line
Other: Acute — The subject will be sited in front of computer screen light illumination for 2 hours.
  Arms: Acute
Other: Chronic — The subject will be sited in front of computer screen light illumination for 2 hours for 5 consecutive days.
  Arms: Chronic

SUMMARY:
The human eye has a dual role, which is reflected by the various photo-receptors used for vision of images and colors ,Image forming photoreceptors (IFP) and for entrainment of our "Biological clock" located in the hypothalamus through the retinal ganglions known as non-image forming photoreceptors (NIFP). The recently discovered new photo-pigment melanopsin which is sensitive to short wavelength (SWL) illumination exists in the-NIFP. The axons of the NIFP form a special nerve known as the Retino-hypothalamic-tract (RHT) that transfers the SWL signal to the biological clock resulting in suppression of pineal melatonin (MLT) production. This is the basic mechanism by which environmental light/dark cycles entrain the biological clock and transfer the message to organs, tissues and cell.

The American Medical Association (AMA) issued a resolution in 2012 stating that light at night constitutes environmental pollution because it violates the daily cycles, including the waking and sleeping cycles, and suppresses the secretion of melatonin from the pineal gland at night. Results of other studies have shown that exposure to artificial light at night (ALAN) and mainly those emerging from SWL sources suppresses MLT-produced in the pineal gland. Computers, tablets, TVs, and smart-phones screens emit SWL illumination, during the day and night hours, whether as active or passive users. The results of previous studies show that, exposure to SWL-ALAN illumination suppresses MLT-secretion and disrupts sleep patterns. In order to understand better the effect of SWL-exposure emerging from screens on human behavior and health, the investigators will study the effects of SWL-exposure on the structure and quality of sleep, cognitive functioning in Continous Performance Test (CPT III), emotional state, and physiological, variables (melatonin secretion levels and body temperature) that were not tested in previous studies.

DETAILED DESCRIPTION:
The investigators will examine whether there is a difference between one-time and multiple exposures to computer screen lighting (350 lux). The investigators hypothesize that multiple and continuous exposure will have a more significant detrimental effect on the quality of sleep and consequently on performance, emotional, and physiological indicators, than one-time exposure to screen light.

Procedure:

On the base-line, first and fifth night of the study, at the end of two hours of exposure to screen light, the subject will be connected to the sleep test system by a skilled technician. On all other nights (nights 2-4), exposure to computer light only, will be conducted and at the end of the exposure the subject will be asked to go to sleep. During the entire experimental period the subject will wear an Actigraph watch to ensure regular sleeping hours. In addition, subjects will be asked not to expose themselves to a computer/tablet/smartphone screen from 20:00 h to wake up.

An Actigraph will monitor their sleep during the week of the experiment. The subject will be invited to attend the Sleep Institute at 21:00 h. The subject will be asked to enter the test room, which will be dark, and sit in front of a computer screen for two hours at a distance of about 60 cm from the screen and perform the on-screen tasks between the hours of 21:00 and 23:00 h. The tasks will include: reading and writing Microsoft Word documents, , and answering questions dealing with a document read and, solving verbal and arithmetic problems, while attempting to accomplish the task correctly and in the quickest time possible. The subject will be told that the purpose of the study is to examine the effect of the content of the tasks on the quality of sleep. During exposure, the subject will be allowed to eat and drink, but do not go to the bathroom. At the end of two hours of exposure to screen light, the subject will be connected to the sleep test system by a skilled technician. Body temperature and 6-hydroxymelatonin sulfate(6-SMT) in the urine will be measured using the on-set and off-set methods three times, at 21:00, 23:00 h, and close to the falling asleep time. Three measurements will be taken after awakening. After the sleep test system is installed, the subject will be asked to go to sleep and in the morning will be woken at his/her average waking time. After the examinee has been woken and has provided a urine sample and body temperature measurement, the sleep test system will be removed and the examinees will be given 30 minutes to organize him/herself, before performing the following tasks to assess his/her degree of fatigue and sleepiness: Continous Performance Test (CPT-III), the Brief Symptoms Inevntory (BSI) emotional questionnaire, and the Epworth Sleepiness Scale (ESS) and Karolinska Sleepiness Scale (KSS) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 20-45,
* healthy
* No history of visual disturbances
* No history of sleep disorders

Exclusion Criteria:

* score more then 5 in the Pittsburgh Questionnaire (PSQI).
* Subjects with a-typicality deviation in the HORNE - OSTBERG sleep-wakefulness cycle questionnaire.
* One of the Eye problems: field of vision, color blindness, or impaired functioning of the pupil in reaction to light.
* Subjects who did shiftwork three months before the experiment
* Subjects that taking sleeping medications in general and melatonin in particular

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
body temperature | 12 hours
  body temperature in celsius degree.physiological marker
Melatonin secretion | 12 hours
  Melatonin -Sulfate Urine ELISA 6-SMT ng/ml. physiological marker
sleepiness | 1 day
  ESS questionnaire score- number
BSI Questionnaire | 1 day
  assess the subject's emotional state- number
Subjective sleepiness | 1 day
  KSS questionnaire-number
attention | 1 hour
  a neuropsychological computerized attention and concentration test, designed to test attentional functions. number
total Sleep time | 1 night
  total sleep time in minutes. physiological marker
Sleep efficiency | 1 night
  percentage of sleep efficiency- physiological marker
sleep latency to sleep stage1 | 1 night
  time in minute to sleep stage 1. physiological marker
sleep latency to sleep stage2 | 1 night
  time in minute to sleep stage 2. physiological marker
wake %TIB | 1 night
  percentage of wake from Time in bed. physiological marker
REM %TIB | 1 night
  percentage of REM from Time in bed. physiological marker
staege1%TIB | 1 night
  percentage of sleep stage1 from Time in bed. physiological marker
stage2%TIB | 1 night
  percentage of sleep stage2 from Time in bed.physiological marker
stage4%TIB | 1 night
  percentage of sleep stage4 from Time in bed.physiological marker

IPD SHARING:
Plan to Share IPD: No